CLINICAL TRIAL: NCT06219629
Title: A Two Part, Observational Basket Study to Determine Usability, Validity and Biomarker Discovery for Mobile EEG, Wearable and Device Collected Objective Measurement of Disturbed Sleep and Neurologic Disorders (LEARNS)
Brief Title: Parkinson's Disease Progression Study
Status: Active, not recruiting | Type: Observational
Sponsor: Koneksa Health (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry); Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: KH007
Record Dates: First submitted 2023-12-04; First posted 2024-01-23 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin biopsies; serum; plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Disease Progression Study

DETAILED DESCRIPTION:
This is a longitudinal, observational Study to Determine Usability, Analytical and Clinical Validity and Biomarker Discovery for Wearable and Mobile Device Collected Objective Measurement of Disturbed Sleep and Neurologic Disorders. The Disease Progression Study part in Parkinson's Disease has a duration of approximately 12 months.

ELIGIBILITY:
Inclusion criteria:

1. Aged ≥18 years to ≤85 years of age.
2. Body mass index (BMI) ≥18 to 40 kg/m2.
3. In adequate health based on medical history and physical examination (other than PD) undertaken following standard care procedures and presenting minimal risk for taking part in the study, per investigator assessment.
4. Participant or caregiver has demonstrated ability to perform satisfactory in-clinic and remote procedures during the screening period.
5. Clinically established PD, consistent with Postuma et al (Mov Disord; 2015).
6. H&Y stage 1 or 2.

Exclusion criteria:

1. Unable to commit to 12 months of data collection.
2. Planning to enroll in a clinical trial for disease modifying therapy that will overlap with the duration of this study.
3. Parkinsonism due to drugs(s) and or toxin(s).
4. Increased risk of falling, defined as >6 falls within the 12 months prior to screening.
5. Urine drug screen positive for opiates, phencyclidine (PCP), cocaine, or amphetamines.
6. Regular binge drinking, defined as ≥4 alcoholic drinks for women or ≥5 alcoholic drinks for men, per investigator assessment.
7. Current or recent (within 6 months prior to screening) diagnosis of a moderate or severe substance use disorder (excluding caffeine) according to Diagnostic and Statistical Manual of Mental Disorders-5 criteria. Note that nicotine use disorder is an exclusion criterion only if it has an effect on sleep (i.e., a participant who routinely awakens at night to smoke), and medical or recreational marijuana is not included in this exclusion criterion.
8. Severe cardiopulmonary, hepatic, renal, or musculoskeletal disease such that activities of daily living are adversely impacted.
9. History of neoplastic disease, with the exception of (1) an adequately treated basal cell carcinoma or carcinoma in situ of the cervix; (2) other malignancies which have been successfully treated >5 years prior to screening without evidence of recurrence.
10. Currently participating in another clinical trial, or previous participation in a clinical trial in which an investigational product was received within 30 days prior to screening or within at least 5 half-lives of the investigational product.
11. Current or planned pregnancy.
12. History of seizures, epilepsy, stroke, multiple sclerosis, or traumatic brain injury (other than mild traumatic brain injury).
13. Intracranial metallic or magnetic devices, such as a cochlear implant or deep brain stimulator.
14. Implanted active device, such as a pacemaker or defibrillator.
15. History of gene therapy, intracranial antisense oligonucleotide treatment, cell transplantation, or experimental brain surgery.
16. Current untreated or unstable depressive disorder or a serious mood disorder requiring hospitalization.
17. Other primary degenerative dementia or neurodegenerative conditions outside of the specific basket in which the participant is enrolled, where applicable.
18. Other uncontrolled infectious, metabolic, or systemic diseases affecting the central nervous system, such as syphilis, hypothyroidism, vitamin B12 or folate deficiency, and other laboratory values.
19. Any other medical, psychiatric, or social condition that, in the opinion of the investigator, is likely to unfavorably alter the risk-benefit of participation, to interfere with protocol compliance, or to confound safety or efficacy assessments.

Additional exclusion criterion for the subset of treatment-naive participants only:

1. No prior treatment to manage motor symptoms of PD; note that brief periods of dopaminergic therapy administered to establish diagnosis are not grounds for exclusion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Compliance; toolkit assessments | Baseline Day 1 through Day 365 End of Participation
  Percentage of total toolkit tasks completed during the remote data collection period

SECONDARY OUTCOMES:
Usability; mobile application | Baseline Day 1 through Day 365 End of Participation
  Percentage of participants reporting a mobile application System Usability Scale (SUS) score ≥68

OTHER OUTCOMES:
Compliance; by category | Baseline Day 1 through Day 365 End of Participation
  Percentage of toolkit assessments completed, by category (motor, speech, and cognitive)
Compliance; by assessment | Baseline Day 1 through Day 365 End of Participation
  Percentage of toolkit assessments completed, by individual assessment
Compliance; wrist-worn device | Baseline Day 1 through Day 365 End of Participation
  Compliance with the wrist-worn device in hours/day
Usability; study phone | Baseline Day 1 through Day 365 End of Participation
  Usability of the study phone, evaluated with the usability questionnaire
Usability; study tablet | Baseline Day 1 through Day 365 End of Participation
  Usability of the study tablet, evaluated with the usability questionnaire
Usability; wrist-worn device | Baseline Day 1 through Day 365 End of Participation
  Usability of the wrist-worn device, evaluated with the usability questionnaire
Usability; software platform | Baseline Day 1 through Day 365 End of Participation
  Usability of the SaaS platform, evaluated with the usability questionnaire
Usable data; toolkit assessments | Baseline Day 1 through Day 365 End of Participation
  Percentage of total toolkit assessments that generate usable data
Usable data; by category | Baseline Day 1 through Day 365 End of Participation
  Percentage of toolkit assessments that generate usable data, by category (motor, speech, and cognitive)
Usable data; by assessment | Baseline Day 1 through Day 365 End of Participation
  Percentage of toolkit assessments that generate usable data, by individual assessment
Usable data; wrist-worn device | Baseline Day 1 through Day 365 End of Participation
  Amount of usable data obtained from the wrist-worn device
Content validity; by assessment | Baseline Day 1 through Day 365 End of Participation
  Content validity evaluated with the in-house content validity survey, by toolkit assessment
Content validity; by PRO | Baseline Day 1 through Day 365 End of Participation
  Content validity evaluated with the in-house content validity survey, by PRO
Criterion validity; toolkit assessments | Baseline Day 1 through Day 365 End of Participation
  Criterion validity evaluated by examining associations between measures derived from the toolkit assessments and disease-specific gold-standard assessments
Criterion validity; wrist-worn device | Baseline Day 1 through Day 365 End of Participation
  Criterion validity evaluated by examining associations between measures derived from the wrist-worn device and disease-specific gold-standard assessments
Construct validity; by data capture location | Baseline Day 1 through Day 365 End of Participation
  Evaluation of the differences between measures obtained remotely versus in-clinic
Construct validity; by data capture frequency | Baseline Day 1 through Day 365 End of Participation
  Evaluation of the differences between measures obtained at different frequencies, such as daily vs weekly
Convergent validity; motor assessments | Baseline Day 1 through Day 365 End of Participation
  Convergent validity evaluated by examining associations between measures derived from the motor assessments
Convergent validity; cognitive assessments | Baseline Day 1 through Day 365 End of Participation
  Convergent validity evaluated by examining associations between measures derived from the cognitive assessments
Convergent validity; speech assessments | Baseline Day 1 through Day 365 End of Participation
  Convergent validity evaluated by examining associations between measures derived from the speech assessments
Discriminant validity; toolkit assessments | Baseline Day 1 through Day 365 End of Participation
  Discriminant validity evaluated by examining associations between measures derived from toolkit assessments identified between categories (motor vs cognitive vs speech)
Evaluation of change; toolkit assessments | Baseline Day 1 through Day 365 End of Participation
  Evaluation of change over time in measures derived from the toolkit assessments
Evaluation of change; wrist-worn device | Baseline Day 1 through Day 365 End of Participation
  Evaluation of change over time in measures derived from the wrist-worn device
Detection of disease progression; toolkit assessments | Baseline Day 1 through Day 365 End of Participation
  Evaluation of change over time in measures derived from the toolkit assessments, comparing progressors and non-progressors as defined by the PGI-C
Detection of disease progression; wrist-worn device | Baseline Day 1 through Day 365 End of Participation
  Evaluation of change over time in measures derived from the wrist-worn device, comparing progressors and non-progressors as defined by the PGI-C
Test-retest reliability; toolkit assessments | Baseline Day 1 through Day 365 End of Participation
  Test-retest reliability evaluated by examining associations between measures derived from the toolkit assessment device captured at adjacent timepoint
Internal consistency reliability; Cronbach's alpha | Baseline Day 1 through Day 365 End of Participation
  Internal consistency reliability evaluated by examining Cronbach's alpha (for composite scores only, as applicable)
Internal consistency reliability; item-total associations | Baseline Day 1 through Day 365 End of Participation
  Internal consistency reliability evaluated by examining item-total associations (for composite scores only, as applicable
Internal consistency reliability; directionality of change | Baseline Day 1 through Day 365 End of Participation
  Internal consistency reliability evaluated by comparing the directionality of change in individual components (for composite scores only, as applicable)
Minimum valid dataset | Baseline Day 1 through Day 365 End of Participation
  Determination of the minimum valid dataset required to monitor disease progression
Comparison of digital and non-digital biomarkers/assessments; toolkit assessments | Baseline Day 1 through Day 365 End of Participation
  Evaluation of the associations between measures derived from the toolkit assessments and non-digital biomarkers
Comparison of digital and non-digital biomarkers/assessments; wrist-worn device | Baseline Day 1 through Day 365 End of Participation
  Evaluation of the associations between measures derived from the wrist-device and non-digital biomarkers
Subgroup analyses | Baseline Day 1 through Day 365 End of Participation
  To evaluate the extent to which compliance, usability, usable data, validity, and reliability differ by subgroup/s
Evaluation of composite scores | Baseline Day 1 through Day 365 End of Participation
  Evaluation of the concepts listed above for composite scores, if applicable

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of Colorado Health Neurosciences Center, Aurora, Colorado
  - Parkinsons Disease And Movement Disorders Center Of Boca Raton, Boca Raton, Florida
  - Accel Research Sites DeLand, DeLand, Florida
  - Accel Research Sites St Petersburg-Largo, Largo, Florida
  - N1 Research LLC, Orlando, Florida
  - Augusta University Health Movement Disorder Clinic, Augusta, Georgia
  - University of Kansas Medical Center Parkinson's Disease and Movement Disorder Center, Kansas City, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Cleveland Clinic, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Upon preliminary analysis (if applicable) and end of study.
Access Criteria: Publications will be shared with Clinical Site Investigators and industry professionals.